CLINICAL TRIAL: NCT06616142
Title: Para-chloro-2-[18F]Fluoroethyl-etomidate ([18F]CETO) as a New PET-tracer for Subtyping in Patients With Primary Aldosteronism - a Pilot Study
Brief Title: Subtyping Primary Aldosteronism With Para-chloro-2-[18F]Fluoroethyl-etomidate
Acronym: SPACE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPACE 2024/176; 2023-508254-26-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Primary Aldosteronism
Keywords: Bilateral adrenal hyperplasia; PET/CT scan; [18F]CETO; Adrenal vein sampling; Primary aldosteronism; Aldosteron producing Adenoma
MeSH Terms: conditions — Hyperaldosteronism | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: All study participants will receive an adrenal vein sampling and a [18F]CETO PET/CT scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aldosterone producing adenoma (Active Comparator): Patients diagnosed with an aldosterone producing adenoma
  Interventions: Drug: [18F]CETO tracer; Drug: Dexamethasone oral; Procedure: Adrenal vein sampling
- Bilateral adrenal hyperplasia (Active Comparator): Patients diagnosed with bilateral adrenal hyperplasia
  Interventions: Drug: [18F]CETO tracer; Drug: Dexamethasone oral; Procedure: Adrenal vein sampling

INTERVENTIONS:
Drug: [18F]CETO tracer — PET/CT with para-chloro-2-[18F]fluoroethyl-etomidate ([18F]CETO) has a high specificity for the steroidogenic enzymes CYP11B1 and CYP11B2, present in the adrenal cortex, and has more favourable tracer characteristics compared to [11C]metomidate. Results obtained with this novel tracer seem promising, but its potential value in the subtyping of PA needs to be further established.
  Other Names: Para-chloro-2-[18F]fluoroethyl-etomidate ([18F]CETO)
Drug: Dexamethasone oral — Pre-treatment of dexamethasone prior to 18F CETO PET/CT scan
Procedure: Adrenal vein sampling — Adrenl vein sampling
  Other Names: AVS

SUMMARY:
The goal of this clinical trial is to investigate the uptake characteristics of [18F]CETO in adrenal tissue in patients with two different subtypes of primary aldosteronism. The main questions it aims to answer are:

* What are the uptake characteristics of [18F]CETO in adrenal tissue in patients with primary aldosteronism?
* What is the concordance between the adrenal vein sampling and the [18F]CETO PET/CT scan results?
* What is the effect of adrenal perfusion on [18F]CETO uptake in the adrenal glands?

Researchers will compare the results of the adrenal vein sampling to a [18F]CETO PET/CT scan to see if the PET/CT can accurately identify the subtypes of primary aldosteronism. Participants will:

* Take dexamethasone three days prior to the scan
* Undergo a [18F]CETO PET/CT
* Report burden of pre-treatment and PET/CT scan

DETAILED DESCRIPTION:
Rationale Primary aldosteronism (PA) is a relatively frequent and clinically relevant secondary cause of hypertension. PA is usually caused by either an aldosterone producing adrenal adenoma (APA) or bilateral adrenal hyperplasia (BAH). Differentiation between these two subtypes is important as it determines the treatment of choice, i.e., unilateral adrenalectomy in case of APA and medical treatment with a mineralocorticoid receptor antagonist in case of BAH. Adrenal vein sampling (AVS) is considered the optimal diagnostic test for this subtyping and is recommended in most patients with PA who are a candidate for surgery. AVS, however, is an invasive and time-consuming procedure with limited availability due to the special expertise required. Additional disadvantages are the risk of procedure related complications and the relative high costs. Thus, there is an unmet need for a non-invasive, faster, more patient friendly and less expensive diagnostic test which can distinguish between the two main subtypes of PA. PET/CT with para-chloro-2-[18F]fluoroethyl-etomidate ([18F]CETO) has a high specificity for the steroidogenic enzymes CYP11B1 and CYP11B2, present in the adrenal cortex, and has more favourable tracer characteristics compared to [11C]metomidate. Results obtained with this novel tracer seem promising, but its potential value in the subtyping of PA needs to be further established. Our hypothesis is that [18F]CETO PET/CT is selectively taken up by aldosterone producing adrenal tissue.

Objective The main objective is to investigate the uptake characteristics of [18F]CETO in adrenal tissue in patients with either APA or BAH. The secondary objective is to evaluate the concordance between the results of adrenal vein sampling and the results of the [18F]CETO scan. In addition, the effect of tissue perfusion on the [18F]CETO uptake by means of a 15O water scan is studied.

Main trial endpoints The main trial endpoint is the investigation of [18F]CETO uptake by adrenal gland tissue in patients with either APA or BAH. Descriptive statistics will be used to explore uptake characteristics.

Secondary trial endpoints The secondary trial end points are i) the concordance between the results of adrenal vein sampling and ii) the relationship between adrenal perfusion and [18F]CETO uptake Trial design Prospective, single-center, diagnostic, observational pilot study. The expected duration of this study is 2 years.

Trial population Adult patients > 18 years of age with biochemically confirmed PA who underwent a successful AVS (n=12) are eligible for inclusion. Main exclusion criteria are diabetes mellitus, serious comorbidity precluding surgery and use of specific medications.

Interventions Participating patients have been subjected to the routine diagnostic work-up for PA as recommended by the guideline of the European Society of Hypertension (2020), including hormonal evaluation before and after a salt-loading protocol, CT or MRI of the adrenal glands and AVS. Three days prior to the PET/CT scans, patients receive pretreatment with dexamethasone in order to enhance tracer specificity. Each participant will be subjected to one additional hospital visit for the investigational diagnostic PET-CT procedure with the administration of [18F]CETO, which is directly preceded by a 15O water scan.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks.

No adverse effects following [18F]CETO and 15O water injection have been reported in the literature. Pretreatment with dexamethasone is recommended for the [18F]CETO PET/CT and could result in mild reversible side effects (hyperglycemia, mood changes, sleep disturbance), which will be monitored by means of a non-invasive questionnaire. As this is a diagnostic pilot study, participating patients will not benefit directly from this investigational diagnostic procedure. However, patients contribute to gathering information on the application of [18F]CETO PET/CT, potentially reducing the need for AVS in future patients.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* Biochemically established diagnosis of PA*
* Completion of standard diagnostic work-up of PA*
* Able to follow and understand instructions to participate in the study
* Able to give written informed consent.

Exclusion Criteria:

* diabetes mellitus (i.e., HbA1c above 42 mmol/mol, and/or fasting plasma glucose > 7.0 mol/l or non-fasting plasma glucose above 11.1 mmol/L )
* serious comorbidities precluding surgery
* severe claustrophobia
* pregnancy/breastfeeding or unable/unwilling to take adequate contraceptives (female only)
* concurrent active infections (e.g., viral, fungal or parasite infections)**
* problematic venous access
* unable/unwilling to take dexamethasone prior to [18F]CETO scanning
* inability to temporary stop medication affecting aldosterone secretion
* use of ketoconazole, metyrapone or cytostatic drugs during previous 6 months***
* long-term use of prednisolone and/or dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Uptake characteristics [18F]CETO | 2 years
  Visual description of uptake characteristics of [18F]CETO uptake in adrenal tissue in patients with APA or BAH.

SECONDARY OUTCOMES:
Concordance adrenal vein sampling and [18F]CETO PET/CT scan | 2 years
  Concordance between the adrenal vein sampling and the results of the [18F]CETO scan will be expressed in percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. M.N. Kerstens, Principal Investigator — Department of Internal Medicine - Endocrinology, University of Groningen, University Medical Center Groningen, Hanzeplein 1, 9713 GZ Groningen, The Netherlands
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing plan has been described in the data management plan.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After end of study.
Access Criteria: Described in the data management plan

REFERENCES:
- [Background] Silins I, Sundin A, Lubberink M, O'Sullivan L, Gurnell M, Aigbirhio F, Brown M, Wall A, Akerstrom T, Roslin S, Hellman P, Antoni G. First-in-human evaluation of [18F]CETO: a novel tracer for adrenocortical tumours. Eur J Nucl Med Mol Imaging. 2023 Jan;50(2):398-409. doi: 10.1007/s00259-022-05957-9. Epub 2022 Sep 8. PMID 36074157
- [Background] Silins I, Sundin A, Nordeman P, Jahan M, Estrada S, Monazzam A, Lubberink M, Aigbirhio F, Hellman P, Antoni G. Para-chloro-2-[18F]fluoroethyl-etomidate: A promising new PET radiotracer for adrenocortical imaging. Int J Med Sci. 2021 Mar 21;18(10):2187-2196. doi: 10.7150/ijms.51206. eCollection 2021. PMID 33859526